CLINICAL TRIAL: NCT07133477
Title: A Randomised, Placebo-Controlled Study to Evaluate the Effect of Fish Oil Concentrate on Skin Function
Brief Title: A Study to Evaluate the Effect of Fish Oil Concentrate on Skin Function
Acronym: NEMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Epax Norway AS (Industry)
Collaborators: Cutest Systems Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AN3991
Record Dates: First submitted 2025-04-22; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Skin Health
Keywords: skin; mono-unsaturated fatty acids; LCMUFA; omega-3

STUDY DESIGN:
Intervention Model Description: Subjects are randomised in a blinded fashion to one of 3 groups. Placebo, dose 1 and dose 2.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will take a total of 4 capsules with a different ratio of fish oil and placebo according to which group they are selected for. Labelling is coded to maintain blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): 1g corn oil capsules
  Interventions: Dietary Supplement: Placebo
- Low dose (Experimental): Subjects will receive 2g of Omega 3-9-11 oil
  Interventions: Dietary Supplement: Omega 3-9-11; Dietary Supplement: Placebo
- High dose (Experimental): Subjects will receive 4g of Omega 3-9-11 oil
  Interventions: Dietary Supplement: Omega 3-9-11

INTERVENTIONS:
Dietary Supplement: Omega 3-9-11 — Fish oil capsules containing a fish oil concentrate from North Atlantic fish species containing EPA / DHA / cetoleic acid and gondoic in controlled amounts.
  Arms: High dose; Low dose
Dietary Supplement: Placebo — Corn oil capsules
  Arms: Low dose; Placebo

SUMMARY:
The primary objective of the study is to determine the benefits of the food product EPAX Omega 3-9-11 on skin function.

Benefits (if any) will be determined by evaluating biophysical measurements of the face and inner forearm. Moreover, the study will determine the dosage effect of Omega-3-9-11 on these measurements.

DETAILED DESCRIPTION:
The long chain mono-unsaturated fatty acids, cetoleic acid (C22:1 n-11) and gondoic acid (C20:1 n-9) found in some North Atlantic fish have been shown to lower inflammatory markers. This has been shown in preclinical studies with particular effect in adipose tissue, and in a human clinical study measuring redness of the face. Omega-3 is also known for reducing skin erythema evoked as a response to UVB exposure, and to decreasing systemic inflammatory biomarkers.

This provides a hypothesis that a combination oil with known bioaccumulation in both subcutaneous fat and in dermal/epidermal layers will contribute to healthy skin function, as shown by a reduction in inflammatory markers and skin erythema and improved barrier function.

The study will recruit subjects to one of 3 arms, a placebo, a low dose and a high dose of omega 3-9-11. Subjects will receive capsules for 3 months and undergo a series of measurements at baseline, 6 weeks and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers who are able to provide signed informed consent
* Healthy male or female volunteers between the ages of 35 and 65 years
* Volunteers with a self-perceived history of atopic skin, prone to redness and/or dryness

Exclusion Criteria:

* Females who are pregnant, breast feeding, or have given birth within the previous 6 weeks or are planning to be pregnant during the study
* Volunteers with previous experience of intolerance or allergic reactions to fish or fish products
* Volunteers with an active skin disorder or a significant history of skin disorders (e.g. psoriasis, eczema, vitiligo, pityriasis versicolor, acne) which in the opinion of a trained assessor or dermatologist may affect the test results
* Volunteers currently taking or who have recently taken antihistamines, antibiotics, systemic anti-inflammatory drugs during the previous week
* Volunteers currently taking or who have recently taken retinoids, immunosuppressive drugs, anti-cancer drugs during the six previous months
* Volunteers who have started, stopped or changed hormonal treatment (including contraceptive pills) in the five previous weeks
* Volunteers whose skin has been exposed to excessive levels of sun or UV rays during the previous month
* Volunteers who are suffering from chronic asthma, a malfunction of the lymphatic system, or an auto immune deficiency disease (e.g. lupus, thyroiditis)
* Volunteers with a history of skin tumours or malignant disease
* Volunteers who have participated in any clinical study involving the test sites within the previous month
* Volunteers taking fish oil supplements or other lipid-based supplements regularly during the last 4 weeks

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Erythema | 3 months intervention
  1. Facial erythema measured using the validated erythema image analysis algorithm within the quantitative measurement system of the Visia CRII image analysis system. Comparison of erythema area (pixels on erythema algorithm map) in pre and post analysis situations will be evaluated statistically for mean and median changes across the study cohort.
Skin hydration | 3 months intervention
  2. Transepithelial water loss will be measured using a non-invasive Tewameter. Values are given as g/m2/hour, higher values relate to increased water loss. Measurements will be made pre and post intervention (for doses together and separately) compared to placebo

SECONDARY OUTCOMES:
Skin parameters, placebo adjusted | 3 months intervention
  1. Facial erythema measured using VISIA facial analysis system and Tewameter, placebo adjusted values between dosing groups.
Skin health by Omega-3 index | 3 months intervention
  4. Primary and secondary measurements as a function of omega-3 index. Omega-3 index is the measurement of EPA and DHA as a % of total lipid in red blood cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Cutest Systems Ltd, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Per patient data will be shared to relevant researchers. All data will be fully anonymised.